CLINICAL TRIAL: NCT05009914
Title: Assessing a New Way of Cardiac Denervation to Reduce the Incidence of Atrial Fibrillation After Coronary Artery Bypass Grafting.
Brief Title: A New Way of Cardiac Denervation to Reduce the Incidence of AF After CABG.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCRC2020003
Record Dates: First submitted 2021-06-29; First posted 2021-08-18 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Denervation; Postoperative Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cardiac denervation group (Experimental): In this group, patients undergoing CABG will receive the procedure of our new way of cardiac denervation, excision of Marshall ligament and Waterstone fat pad.
  Interventions: Procedure: cardiac denervation
- controlled group (No Intervention): In this group ,patients undergoing CABG will not receive the procedure of cardiac denervation.

INTERVENTIONS:
Procedure: cardiac denervation — Excision of Marshall ligament and Waterstone fat pad during CABG.
  Arms: cardiac denervation group

SUMMARY:
This is a prospective, random controlled trial(RCT) study. 430 patients undergoing coronary artery bypass grafting were enrolled. Our new way of cardiac denervation, defined as excision of Marshall ligament and Waterstone fat pad, was performed in 215 patients, and the other 215 patients were used as control subjects. All the patients need to equip with electronic monitor to record heart rhythms within 6 days after CABG. The investigators will compare the incidence of postoperative atrial fibrillation between two groups, and follow up 30 days after discharged.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing simple CABG (on-pump/off-pump) for the first time.
2. Patients who signed the informed consent form and willing to undergo cardiac denervation.

Exclusion Criteria:

1. Age < 18；
2. Emergent CABG;
3. Cardiac surgery history；
4. Receiving other cardiac surgery except of CABG at the same time, such as Morrow、valvular surgery、ventricular aneurysm surgery、congenital heart diseases surgery；
5. Requiring mechanical or pharmacological therapy for hemodynamic support before CABG, such as ECMO or IABP;
6. History of AF ;
7. Taking antiarrhythmic agents except of beta-blockers last 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of POAF during hospital. | 6 days after surgery.
  Incidence of postoperative atrial fibrillation after surgery during hospital.

SECONDARY OUTCOMES:
Incidence of massive haemorrhage needing blood transfusion caused by cardiac denervation. | Postoperative hospitalization, an average of 8 days.
  The incidence of massive haemorrhage needing blood transfusion caused by cardiac denervation during in-hospital time.
Incidence of transferring to on-pump CABG caused by cardiac denervation. | Intraoperatively.
  The incidence of transferring to on-pump CABG caused by cardiac denervation during in-hospital time.
Incidence of re-operation aiming to stop bleeding caused by cardiac denervation. | Postoperative hospitalization, an average of 8 days.
  The incidence of re-operation aiming to stop bleeding caused by cardiac denervation during in-hospital time.
Incidence of pericarial effusion within 30 days after discharged. | within 30 days after discharged.
  The incidence of pericarial effusion within 30 days after discharged.
Incidence of arrhythmia exclude of AF within 30 days after discharged. | within 30 days after discharged.
  The incidence of arrhythmia exclude of AF within 30 days after discharged.
Postoperative length of hospitalization. | Postoperative hospitalization, an average of 8 days.
  Each participant's oostoperative length of hospitalization.
All cost after surgery. | Postoperative hospitalization, an average of 8 days.
  All cost associated with treatment after surgery during in-hospital time.
MACCE | within 30 days after discharged.
  major adverse cardiovascular and cerebrovascular events (MACCE), which was defined as the composite of stroke, myocardial infarction, repeat coronary revascularization and all-cause mortality during the 30-day follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Feng, MD PhD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Z, Tiemuerniyazi X, Xu F, Wang Y, Sun Y, Yan P, Tian L, Han C, Zhang Y, Pan S, Hu Z, Li X, Zhao W, Feng W. Partial Cardiac Denervation to Prevent Postoperative Atrial Fibrillation After Coronary Artery Bypass Grafting: The pCAD-POAF Randomized Clinical Trial. JAMA Cardiol. 2025 Jan 1;10(1):71-77. doi: 10.1001/jamacardio.2024.4639. PMID 39550720